CLINICAL TRIAL: NCT04156009
Title: Aromatherapy for Procedural Anxiety in Pain Management and Interventional Spine Procedures
Brief Title: Lavender Aromatherapy Spine Procedure Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 19-06020284
Record Dates: First submitted 2019-11-01; First posted 2019-11-07 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Spine Injuries and Disorders; Pain, Back
Keywords: aromatherapy; lavender; anxiety; spine intervention
MeSH Terms: conditions — Disease; Back Pain; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Masking Description: For the treatment group, the aromatherapy tablets will be activated for max aromatherapy. For the control group, the tablets will not be activated and will be devoid of scent. For both groups, the tablet will be wrapped in masking tape to maintain the blind for subjects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (+aromatherapy) group (Experimental)
  Interventions: Other: Activated Lavender Elequil aromatabs® (#372)
- Control (-aromatherapy) group (Sham Comparator)
  Interventions: Other: Unactivated Lavender Elequil aromatabs® (#372)

INTERVENTIONS:
Other: Activated Lavender Elequil aromatabs® (#372) — Activated Lavender aromatherapy tablets wrapped in tape
  Arms: Treatment (+aromatherapy) group
Other: Unactivated Lavender Elequil aromatabs® (#372) — Unactivated Lavender aromatherapy tablets wrapped in tape
  Arms: Control (-aromatherapy) group

SUMMARY:
Patient anxiety prior to invasive procedures poses a significant barrier to successful treatment if not well-managed. The purpose of this study is to evaluate lavender aromatherapy, a non-sedating alternative, to reduce anxiety prior to interventional spinal procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females between 18-85 years old
2. Scheduled for one of the following procedures on the day of consent:

   1. Epidural steroid injection (ESI)
   2. Medial branch block (MBB)
   3. Radiofrequency ablation (RFA)
3. Able to provide informed consent

Exclusion Criteria:

1. History of anxiety disorder
2. Currently on anxiolytic therapy
3. Poor sense of smell
4. Allergy/aversion to aromatherapy
5. Non-English speaking

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2020-01-29 (Actual); Primary Completion 2020-11-18 (Actual); Study Completion 2020-11-18 (Actual)

PRIMARY OUTCOMES:
Change in Subjects' Anxiety State as measured by the State Trait Anxiety Inventory (STAI-6) | Administered within 30 minutes before and 30 minutes after intervention
  The STAI-6 is a six-item assessment of state anxiety. Each item is assessed on a four-point Likert scale. Scores on the STAI-6 range from 6-24, with a higher score indicating greater state anxiety.

SECONDARY OUTCOMES:
Number of Vasovagal Events during Standard of Care Spine Procedure | Assessed within 30 minutes following the standard of care spine procedure
  All vasovagal events that occur during the standard of care spine procedure will be recorded and reported
Number of Aborted Standard of Care Spine Procedures | Assessed within 30 minutes following standard of care spine procedure completion or abortion

CONTACTS AND LOCATIONS:
Overall Officials: Jaspal R Singh, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal to achieve aims in the approved proposal.